CLINICAL TRIAL: NCT02946879
Title: Long-term Follow-up Study of Participants Following an Open Label, Multi-centre, Phase I/II Dose Escalation Trial of an Adeno-associated Virus Vector (AAV2/5-OPTIRPE65) for Gene Therapy of Adults and Children With Retinal Dystrophy Owing to Defects in RPE65 (LCA2)
Brief Title: Long-Term Follow-Up Gene Therapy Study for Leber Congenital Amaurosis OPTIRPE65 (Retinal Dystrophy Associated With Defects in RPE65)
Status: Completed | Type: Observational
Sponsor: MeiraGTx UK II Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT004; 2016-000898-20 (EudraCT Number)
Record Dates: First submitted 2016-07-22; First posted 2016-10-27 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Leber Congenital Amaurosis (LCA); Eye Diseases; Eye Diseases, Hereditary; Retinal Diseases
MeSH Terms: conditions — Leber Congenital Amaurosis; Eye Diseases; Eye Diseases, Hereditary; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Low dose AAV OPTIRPE65: subretinal administration of a single low dose of AAV RPE65
  Interventions: Biological: AAV OPTIRPE65
- Intermediate dose AAV OPTIRPE65: subretinal administration of a single intermediate dose of AAV RPE65
  Interventions: Biological: AAV OPTIRPE65
- High dose AAV OPTIRPE65: subretinal administration of a single highdose of AAV RPE65
  Interventions: Biological: AAV OPTIRPE65

INTERVENTIONS:
Biological: AAV OPTIRPE65 — comparison of different doses of AAV RPE65

SUMMARY:
This study is a longer-term follow-up study for patients who have been administered AAV2/5-OPTIRPE65 in the Phase I/II, open label, non-randomised, two-centre, dose escalation trial in adults and children with retinal dystrophy associated with defects in RPE65.

DETAILED DESCRIPTION:
The follow up study is designed to collect data on longer-term safety and efficacy of AAV2/5-OPTIRPE65 administration in the OPTIRPE65 trial.

ELIGIBILITY:
Inclusion Criteria:

* Were enrolled and treated in the prior open-label, Phase I/II, dose escalation study involving intraocular administration of AAV2/5-OPTIRPE65

Exclusion Criteria:

* Individuals will be excluded if they are unwilling or unable to meet with the requirements of the study.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population are those with Leber Congenital Amaurosis (LCA) with gene mutation RPE65 who have participated in the OPTIRPE65 trial.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-11; Primary Completion 2023-07 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events related to the treatment | 5 years
  Safety is defined as the absence of ATIMP-related safety events

SECONDARY OUTCOMES:
Improvement in the retinal function | 5 years
  Improvements in visual function as assessed by visual assessment
Improvement in the visual function | 5 years
  Improvements in retinal function as assessed by visual assessment
Improvement in quality of life | 5 years
  Improvement in the participant's quality of life which is measurable by QoL questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Kellogg Eye Center, University of Michigan Health, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided